CLINICAL TRIAL: NCT03822533
Title: A Cost-efficiency Analysis of Physiotherapist or Physicians as Primary Assessors for Patients With Knee Pain in Primary Care
Brief Title: A Cost-efficiency Analysis of Primary Assessors for Patients With Knee Pain in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 115841healthecon
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Primary assessor; cost efficiency; physiotherapist; quality of life
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapists; Physicians

STUDY DESIGN:
Intervention Model Description: Participants with suspected knee osteoarthritis are either randomised to a physiotherapist or a physician as primary assessor for assessment and treatment. After the first assessment that the patients are assigned to, the patients can choose to seek the other health care provider if they want to.
  This study focuses on analysing cost efficiency of the health care processes for patients with suspected knee osteoarthritis in primary care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapist as primary assessor (Other): The healthcare process will be started with a physiotherapist assessment and treatment. Treatments could involve individual or group treatment including patient education and physical exercise.
  Patients can seek a physician anytime after the first assessment with the physiotherapist.
  Interventions: Other: Physiotherapist as primary assessor
- Physician as primary assessor (Other): The healthcare process will be started with a physician assessment and treatment. Treatments could involve drug prescription, referral to x-ray, referral to other healthcare providers and sick-leave.
  Patients can seek a physiotherapist anytime after the first assessment with the physician.
  Interventions: Other: Physician as primary assessor

INTERVENTIONS:
Other: Physiotherapist as primary assessor — Physiotherapist diagnose and treat the patient.
  Arms: Physiotherapist as primary assessor
Other: Physician as primary assessor — Physician diagnose and treat the patient.
  Arms: Physician as primary assessor

SUMMARY:
Background: Almost half of the Swedish population are overweight or obese. This will probably affect the incidence of osteoarthritis since overweight is a strong risk factor. Osteoarthritis consultations is expected to increase with 30-50% within the next 20 years. Today, in Swedish primary care, both physicians and physiotherapists are primary assessors for patients with suspected knee osteoarthritis. A task shifting with physiotherapists as the only primary assessor could increase the access rate to physicians in primary care for patients with more severe disorders. Yet, it is unclear what effects these different healthcare processes have and the costs of it.

Purpose: The overall purpose of this study is to perform an economic evaluation of two healthcare processes, where a healthcare process initiated by a physiotherapist is compared with when it is initiated with a physician for patients with suspected knee osteoarthritis.

Methods: 100 patients will be randomized either to a physiotherapists or to a physician for first assessment, diagnosis and treatment. Measurements of health-related quality of life and costs for visits to physiotherapists, physician or other healthcare provider, drug prescriptions and sick-leave will be collected. A cost-effectiveness analysis will be conducted, presenting incremental cost-effectiveness ratio (ICER) and a non-parametric bootstrapping will be conducted to demonstrate the uncertainties surrounding the ICER.

Expected results: It is expected that this randomized controlled study will show the effects on quality adjusted life years, cost-efficiency and cost-utility of two different primary assessors for patients with suspected knee osteoarthritis consulting primary care. The results could clarify which profession that is most appropriate to be the primary assessor for patients with suspected knee osteoarthritis in primary care.

DETAILED DESCRIPTION:
Problem statements:

What is the difference in cost efficiency between a healthcare process with a physiotherapists as primary assessor and a physician as primary assessor for patients with suspected knee osteoarthritis?

Which effect does a clinical pathway with a physiotherapists as primary assessor for patients with suspected knee osteoarthritis have on quality adjusted life years compared with a physician as primary assessor?

What are the differences in costs between the two healthcare processes initiated by either a physiotherapist or a physician set against the differences in effects?

Patient recruitment:

Some data has already been collected for another clinical trial (ID: NCT03715764), which will be used in this study too. The patient recruitment is finished, while data collection regarding cost variables has not started yet.

Patients were recruited from primary care centers and rehabilitation centers in southwestern Sweden.

Screening procedure:

Nurses and administration personnel at the recruitment units got information about the study and the screening protocol from the data collector and project leader. Each recruiting unit had a contact person that were responsible for the protocols and to contact the data collector when an eligible patient was found. It was regular contact between the project leader and the contact persons at the recruiting units. All screening protocols were sent to the data collector. All participants got orally and written information about the study from the data collector, and patients provided written informed consent.

Randomization:

A computer-generated list of random numbers was used, where participants were randomly assigned to being assessed, diagnosed and treated either by a physiotherapist or a physician first. The project coordinator managed the sequence generation, allocation concealment, enrolment and assignments of participants and kept the concealed randomization scheme and sequentially numbered, sealed envelopes in a locked cupboard (in the same building where the enrolment was), only available for the project coordinator. The project coordinator revealed the allocation to the participant shortly after the baseline measurement and to the health care providers. Data collector, data analyst and statistician were blinded of allocation until completion of data collection for the primary outcome measures at the 12 months follow up for the last recruited patient. Group allocation was revealed when analysing data for the other clinical trial (ID: NCT03715764).

The project coordinator was not involved in the screening procedure nor the data collection, and was not included among the healthcare providers in the study. The blinded data collector and analyst, whom is a physiotherapists, were not involved in assessing, diagnosing and treating patients with knee osteoarthritis while the first study (ID: NCT03715764) was conducted.

Data collection:

Demographic data and measurements of health-related quality of life (HrQoL) has already been collected for another clinical trial (ID: NCT03715764). These data will also be used for the cost-efficiency analysis. Demographic data were collected at baseline. Measurements of HrQoL were measured with EuroQol 5 dimensions 3 levels (EQ5D-3L) and collected at baseline (before randomization), 3- , 6- and 12 months follow ups.

New data collection will be made for cost variables. Data regarding costs for the healthcare processes will be extracted from patient journals. The costs for visits to physiotherapists, physician or other healthcare providers will be collected from the healthcare organization. The drug prices will be collected from the Swedish Association of Local Authorities and Regions for the time period the drugs were prescribed. Production loss due to sick-leave and health care visits will be valued according to mean gross salary (including taxes and social fees).

Calculating total costs (number of contacts per patient * costs ) for:

* Physiotherapy contacts in primary care
* Physician contacts in primary care
* Referrals to x-ray
* Referrals to other healthcare givers
* Drug prescriptions
* Sick-leave days

Data management:

All data will be coded and managed according to the General Data Protection Regulation. All data will be confidential and only authorized will have access to the patient registry. No individual information can be identified since the results will be presented at group level. Data will be saved for at least 10 years to enable audit.

Sample size:

A sample size of 50 patients per group will be necessary to detect a minimal clinical improvement of 0.121(SD 0.2) on the EQ5D-3L-index, given an anticipated dropout rate of 14%. The sample size calculation was calculated with a two-sided 5% significance level and a power of 80%.

Statistical analysis plan:

Data will be analyzed descriptively and presented as numbers and percent, mean and standard deviation or median and 25th to 75th percentiles. Statistical analysis will be made in SPSS Windows and the analysis will be applied with intention-to-treat (ITT).

The economic evaluation will be developed together with a health economist. The method will be a cost-effectiveness analysis alongside the clinical trial comparing costs and effects for the two alternatives based on collected data from the trial. The EQ5D-3L measurements will be used for analyzing quality adjusted life years. The result will be presented as an incremental cost-effectiveness ratio (ICER) and a non-parametric bootstrapping will be conducted to demonstrate the uncertainties surrounding the ICER.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain most of the days the last month
* Over 38 years old
* Crepitus on active motion
* Morning stiffness less than 30 minutes

Exclusion Criteria:

* Not been diagnosed for current knee pain
* Non-traumatic cause due to current knee pain
* No other rheumatic, severe somatic or psychological diseases that can affect the outcome measures.
* Not pregnant
* Does not know enough Swedish to answer questionnaires.

Min Age: 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2022-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lena Nordeman, PhD, Principal Investigator — Närhälsan Research and development center Södra Älvsborg
Locations (9):
- Sweden (9):
  - Närhälsan Vänersborg Rehabmottagning, Vänersborg, VastraGotaland
  - Medpro Clinic Brålanda-Torpa Vårdcentral, Brålanda, Västra Götaland County
  - Medpro Clinic Lilla Edet Vårdcentral, Lilla Edet, Västra Götaland County
  - Närhälsan Lilla Edets Rehabmottagning, Lilla Edet, Västra Götaland County
  - Capio Läkarhus Hjortmossen, Trollhättan, Västra Götaland County
  - Närhälsan Trollhättan Rehabmottagning, Trollhättan, Västra Götaland County
  - Primapraktiken, Trollhättan, Västra Götaland County
  - Medpro Clinic Torpa Vårdcentral, Vänersborg, Västra Götaland County
  - Vårdcentralen Nordstan, Vänersborg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turkiewicz A, Petersson IF, Bjork J, Hawker G, Dahlberg LE, Lohmander LS, Englund M. Current and future impact of osteoarthritis on health care: a population-based study with projections to year 2032. Osteoarthritis Cartilage. 2014 Nov;22(11):1826-32. doi: 10.1016/j.joca.2014.07.015. Epub 2014 Jul 30. PMID 25084132
- [Background] Walters SJ, Brazier JE. Comparison of the minimally important difference for two health state utility measures: EQ-5D and SF-6D. Qual Life Res. 2005 Aug;14(6):1523-32. doi: 10.1007/s11136-004-7713-0. PMID 16110932
- [Background] Brazier JE, Harper R, Munro J, Walters SJ, Snaith ML. Generic and condition-specific outcome measures for people with osteoarthritis of the knee. Rheumatology (Oxford). 1999 Sep;38(9):870-7. doi: 10.1093/rheumatology/38.9.870. PMID 10515649
- [Derived] Ho-Henriksson CM, Svensson M, Thorstensson CA, Nordeman L. Physiotherapist or physician as primary assessor for patients with suspected knee osteoarthritis in primary care - a cost-effectiveness analysis of a pragmatic trial. BMC Musculoskelet Disord. 2022 Mar 17;23(1):260. doi: 10.1186/s12891-022-05201-3. PMID 35300671

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (n=294)
  * Not meeting inclusion criteria (n=185)
  * Declined to participate (n=15)
  * Excluded due to exclusion criteria (n=94)
Groups:
- Physiotherapist as Primary Assessor: The healthcare process started with a physiotherapist assessment and treatment. Treatments could involve individual or group treatment including patient education and physical exercise.
  Patients could seek a physician anytime after the first assessment with the physiotherapist.
  Physiotherapist as primary assessor: Physiotherapist diagnosed and treated the patient.
- Physician as Primary Assessor: The healthcare process started with a physician assessment and treatment. Treatments could involve drug prescription, referral to x-ray, referrals to other healthcare providers and sick-leave.
  Patients could seek a physiotherapist anytime after the first assessment with the physician.
  Physician as primary assessor: Physician diagnosed and treated the patient.
Period: Baseline
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Started | 35 | 34
Completed | 35 | 34
Not Completed | 0 | 0
Period: 3 Month Follow-up
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Started | 35 | 34
Completed | 30 | 28
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 2 | 2
Period: 6 Month Follow-up
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Started | 30 | 28
Completed | 27 | 28
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0
Period: 12 Month Follow-up
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Started | 27 | 28
Completed | 21 | 23
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Surgery | 2 | 0
Not completed — Wrong address | 1 | 0
Not completed — No symptoms | 1 | 0
Not completed — Changed primary care center | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Physician as Primary Assessor: The healthcare process started with a physician assessment and treatment. Treatments could involve drug prescriptions, referral to x-ray, referrals to other healthcare providers and sick-leave.
  Patients could seek a physiotherapist anytime after the first assessment with the physician.
  Physician as primary assessor: Physician diagnosed and treated the patient.
- Total: Total of all reporting groups
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (12) | 59 (12) | 60 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 14 | 11 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Level of education [Count of Participants; unit: Participants]
  Primary school | 8 | 4 | 12
  Secondary school | 15 | 20 | 35
  Tertiary school | 12 | 10 | 22
Current Employment [Count of Participants; unit: Participants]
  Employed/working | 19 | 18 | 37
  Unemployed | 0 | 1 | 1
  Retired/early retirement | 15 | 13 | 28
  Sick leave | 1 | 2 | 3
Pain duration (months) [Mean (Standard Deviation); unit: months] | 14 (22) | 10 (16) | 12 (19)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30 (4.4) | 29 (6.7) | 29 (5.6)
Health-related quality of life [Mean (Standard Deviation); unit: score on a scale] — Health-related quality of life was used as the generic measure for health improvement and was measured at baseline, 3-, 6- and 12-month follow-up. The Swedish version of Euroqol-5 dimensions-3 levels (EQ5D-3L) was used to assess perceived self-rated health-related quality of life. The questionnaire contained five dimensions and resulted in an index ranging from -0,549 to 1 using the United Kingdom tariffs. An index of 1 indicate full health. Only the baseline value is presented. The index was collected to calculate quality adjusted life years (QALY), see Primary outcome.
  score on a scale | 0.73 (0.121) | 0.62 (0.222) | 0.67 (0.185)
Pain intensity (visual analogue scale 0-100) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity were collected using a visual analogue scale (VAS) ranging from 0 to 100, were 0 represents no pain and 100 worst imaginable pain.
  units on a scale | 45 (15.9) | 52 (16.4) | 49 (16.5)
Physical function in lower extremities [Mean (Standard Deviation); unit: number of stands from sitting on a chair] — Physical function were measured with the performance test, 30 seconds chair stand test, where patients were encouraged to perform as many stands as possible in 30 seconds. The start position was sitting on a chair. The stands were counted if the participant were fully raised to straight hips and knees. The arms were folded across the chest during the test.
  number of stands from sitting on a chair | 12 (4.6) | 11 (3.3) | 12 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Quality Adjusted Life Years (QALY)
Description: Health-related quality of life was used as the generic measure for health improvement and was measured at baseline, 3-, 6- and 12-month follow-up. The Swedish version of Euroqol-5 dimensions-3 levels (EQ5D-3L) was used to assess perceived self-rated health-related quality of life. The questionnaire contained five dimensions and resulted in an index ranging from -0,549 to 1 using the United Kingdom tariffs. An index of 1 indicate full health. For each participant, EQ-5D-3L index was used when calculating quality adjusted life years (QALY) using linear interpolation between each measurement point and the trapezoidal rule to calculate the "area under the curve". QALY range from 0 to 1, where 0 means death and 1 equals full health.
Time Frame: 12 months
Population: Total 21 patients participated in the 12 month follow up in the physiotherapy group and 23 in the physician group. Imputation using multiple imputation and the analysis included all enrolled patients in each group (35 in the physiotherapy group, and 34 in the physician group).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Number analyzed (Participants) | 35 | 34
score on a scale | 0.74 (0.17) | 0.73 (0.18)
Statistical Analysis 1: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Mean difference using independent samples t-test; Test type: Superiority; p = 0.69, t-test, 2 sided; Mean Difference (Final Values) = 0.015, 95% CI 2-sided [-0.059 to 0.089]
Statistical Analysis 2: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Presenting β-values from linear regression analysis for group variable adjusted for baseline differences in EQ-5D-3L-index. The results from this analysis were used to calculate incremental cost-effectiveness ratio (mean difference in costs divided by mean difference in QALYs); Test type: Superiority; Regression, Linear — The linear regression analysis was needed to calculate the incremental cost efficiency ratio (ICER). The p-value from this test was not relevant for the ICER calculation; First step in a cost-efficiency analysis; Mean Difference (Final Values) = -0.015, 95% CI 2-sided [-0.093 to 0.063]

2. Primary Outcome: Mean Difference in Total Costs (Societal Perspective)
Description: Total costs with the societal perspective includes health care visits, prescribed drugs, productivity loss and unpaid work compensation. Data were retrieved from medical records.
Time Frame: 12 months
Population: Based on retrieved medical records where 32 patients could be analysed in the physiotherapy group and 29 patients in the physician group regardless if they attended to the planned follow ups in the study.
Measure: Mean (Standard Deviation); unit: Euro (currency)
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Number analyzed (Participants) | 32 | 29
Euro (currency) | 633 (620) | 996 (1276)
Statistical Analysis 1: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Independent-samples t-test. Dependent variable cost items, independent variable group (physiotherapist or physician assessment); Test type: Superiority; p = 0.17, t-test, 2 sided; Mean Difference (Final Values) = -364, 95% CI 2-sided [-891 to 164]
Statistical Analysis 2: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Test type: Superiority; Regression, Linear — [p-value comment as in outcome 1, analysis 2]; First step in a cost-efficiency analysis; Mean Difference (Final Values) = -364, 95% CI 2-sided [-870 to 143]

3. Primary Outcome: Mean Difference in Total Costs (Health Care Perspective)
Description: Health care perspective includes health care visits and prescribed drugs. Data were collected through medical records.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Euro (currency)
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Number analyzed (Participants) | 32 | 29
Euro (currency) | 515 (541) | 748 (885)
Statistical Analysis 1: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.23, t-test, 2 sided; Mean Difference (Final Values) = -233, 95% CI 2-sided [-616 to 150]
Statistical Analysis 2: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Linear regression analysis. The results from this analysis were used to calculate incremental cost-effectiveness ratio (mean difference in costs divided by mean difference in QALYs); Test type: Superiority; Regression, Linear — [p-value comment as in outcome 1, analysis 2]; First step in a cost-efficiency analysis; Mean Difference (Final Values) = -233, 95% CI 2-sided [-605 to 139]

4. Primary Outcome: Incremental Cost-effectiveness Ratio (ICER) - Societal Perspective
Description: Mean difference in costs divided by mean difference in quality adjusted life years (QALYs). Presenting the results of the cost-effectiveness analysis (ICER). Societal perspective includes health care visits, prescribed drugs, productivity loss and unpaid work compensation
  Incremental Cost-effectiveness Ratio was derived from the model where a measure of dispersion was not an output of the model
Time Frame: 12 months
Population: All enrolled patients were included in this analysis which included imputed data.
Measure: Number; unit: Ratio (Euro/QALY)
Groups:
- Physiotherapy Assessment vs Physician Assessment: Physiotherapy assessments costs and effects on quality adjusted life years were compared to the costs and effects of physician assessment.
Arm/Group | Physiotherapy Assessment vs Physician Assessment
Number analyzed (Participants) | 69
Ratio (Euro/QALY) | 24266

5. Primary Outcome: Incremental Cost-effectiveness Ratio (ICER) - Health Care Perspective
Description: Mean difference in costs divided by mean difference in quality adjusted life years (QALYs). Presenting the results of the cost-effectiveness analysis (ICER). Health care perspective includes health care visits and prescribed drugs.
  Incremental Cost-effectiveness Ratio was derived from the model where a measure of dispersion was not an output of the model
Time Frame: 12 months
Population: All enrolled patients were included in this analysis which included imputed data.
Measure: Number; unit: Ratio (Euro/QALY)
Groups:
- Physiotherapy vs Physician as Primary Assessors: Physiotherapy assessments costs and effects on quality adjusted life years were compared to the costs and effects of physician assessment.
Arm/Group | Physiotherapy vs Physician as Primary Assessors
Number analyzed (Participants) | 69
Ratio (Euro/QALY) | 15533

6. Secondary Outcome: Costs for Physiotherapy Visits
Description: Number of visits registered in patients journal multiplied with the cost.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Euro (currency)
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Number analyzed (Participants) | 32 | 29
Euro (currency) | 380 (377) | 332 (641)
Statistical Analysis 1: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Test type: Superiority; p = 0.72, t-test, 2 sided; Mean Difference (Final Values) = 48, 95% CI 2-sided [-219 to 314]

7. Secondary Outcome: Costs for Physician Visits
Description: Number of visits registered in patients journal multiplied with cost
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Euro (currency)
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Number analyzed (Participants) | 32 | 29
Euro (currency) | 39 (95) | 217 (140)
Statistical Analysis 1: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Test type: Superiority; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = -178, 95% CI 2-sided [-239 to 118]

8. Secondary Outcome: Costs for Referrals to Radiography
Description: Number of referrals to radiography registered in patients journal multiplied with its costs
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Euro (currency)
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Number analyzed (Participants) | 32 | 29
Euro (currency) | 7.9 (25) | 32 (42)
Statistical Analysis 1: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Final Values) = -24, 95% CI 2-sided [-42 to 6.2]

9. Secondary Outcome: Costs for Referrals to Orthopedic Surgeon
Description: Number of referrals to orthopedic surgeon registered in patients journal multiplied with the costs
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Euro (currency)
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Number analyzed (Participants) | 32 | 29
Euro (currency) | 22 (85) | 33 (100)
Statistical Analysis 1: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Test type: Superiority; p = 0.62, t-test, 2 sided; Mean Difference (Final Values) = -12, 95% CI 2-sided [-59 to 36]

10. Secondary Outcome: Costs for Collected Prescribed Drugs
Description: Data extraction from a drug database for prescribed drugs belonging to the Anatomical Therapeutic Chemical Classification groups M01 anti-inflammatory and anti-rheumatic products, M02 topical products for joint and muscular pain, M03 muscle relaxants, M09 other drugs for disorders of the musculoskeletal system, N02A opioids, N02B other analgesics and antipyretics.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Euro (currency)
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Number analyzed (Participants) | 32 | 29
Euro (currency) | 7.8 (34) | 6.6 (16)
Statistical Analysis 1: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Test type: Superiority; p = 0.87, t-test, 2 sided; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-13 to 15]

11. Secondary Outcome: Costs for Productivity Loss
Description: Productivity loss included the time for visiting health care, telephone calls, traveling, waiting time and costs for sick leave days. The costs was calculated with gross salary including social fees.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Euro (currency)
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Number analyzed (Participants) | 32 | 29
Euro (currency) | 111 (91) | 365 (853)
Statistical Analysis 1: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Test type: Superiority; p = 0.27, t-test, 2 sided; Mean Difference (Final Values) = -254, 95% CI 2-sided [-728 to 220]

12. Secondary Outcome: Costs for Unpaid Work Compensation
Description: The costs for the time the patients were visiting health care or consulting via telephone, including traveling and waiting time. Production loss was calculated with net mean salary. Included participants that reported they were retired or unemployed.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Euro (currency)
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
Number analyzed (Participants) | 32 | 29
Euro (currency) | 125 (103) | 123 (191)
Statistical Analysis 1: Comparison: Physiotherapist as Primary Assessor vs Physician as Primary Assessor; Test type: Superiority; p = 0.96, t-test, 2 sided; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-113 to 118]

ADVERSE EVENTS:
Time Frame: 1 year from baseline
Arm/Group | Physiotherapist as Primary Assessor | Physician as Primary Assessor
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

LIMITATIONS AND CAVEATS:
Major organizational changes in Vastra Gotaland Region, where the study was conducted, affected the recruiting process. The research project was probably de-prioritized since the patient flow declined drastically. Hence the target number of participants needed to achieve target power was not reached due to early termination of the recruiting process.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03822533/Prot_SAP_000.pdf